CLINICAL TRIAL: NCT00165516
Title: A Phase II Feasibility Study of Extrapleural Pneumonectomy With Intraoperative Intrathoracic/Intraperitoneal Heated Cisplatin With Amifostine and Sodium Thiosulfate
Brief Title: Extrapleural Pneumonectomy With Intraoperative Intrathoracic/Intraperitoneal Heated Cisplatin With Amifostine and Sodium Thiosulfate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-302
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Pleural Mesothelioma; Malignant Pleural Mesothelioma
Keywords: Extrapleural pneumonectomy; cisplatin; heated cisplatin
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Cisplatin; sodium thiosulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cisplatin — Heated and given as an one-hour lavage of the chest and abdomen during surgery
Drug: Sodium Thiosulfate — After the one-hour lavage, sodium thiosulfate is given intravenously

SUMMARY:
The purposes of this study are: to evaluate the effects (good and bad) that administering heated cisplatin into the chest and abdomen cavity following surgical resection has on malignant mesothelioma; to collect data on the toxicity of cisplatin given directly into the chest and abdomen, and the levels of the cisplatin in the body; to determine if this treatment method has the possibility of helping patients with pleural mesothelioma live longer; and to determine if this treatment method can help decrease the rate of local recurrence of mesothelioma.

DETAILED DESCRIPTION:
* Patients will undergo surgery called extrapleural pneumonectomy which involves removal of the lung, the lining of the lung, the covering of the heart, and the muscle that separates the chest and abdomen. At the conclusion of the resection, if the patient has less then 1 cm3 of residual gross disease in one or more areas, then the heated chemotherapy lavage will begin. If more than this volume of disease is present, then the patient will receive additional treatment off-study.
* The chemotherapy treatment consists of a one-hour lavage of the chest and abdomen cavity with heated cisplatin given in the operating room through the surgical incision. At the completion of the hour, sodium thiosulfate is given intravenously to reduce the potential side effects of cisplatin.
* During the surgery and for four hours following the completion of the cisplatin lavage, blood samples, urine samples, chest wall muscle samples, and samples of the chemotherapy solution will be done in order to measure the concentration of chemotherapy and the impact of cisplatin on the various cell samples.
* Patients will remain in the hospital until they have recovered from surgery (7-14 days). Following discharge from the hospital, patients will be seen 1-2 weeks post-operatively for blood tests. 6 weeks later additional blood tests and and echocardiogram will be performed. This echocardiogram will be repeated 6 months post-operatively to re-assess heart function.

ELIGIBILITY:
Inclusion Criteria:

* Male of non-pregnant female 18 years of age or older
* HIstopathologic confirmation of malignant pleural mesothelioma
* Ejection fraction > 45%
* Evidence of adequate renal and hepatic function
* Grossly normal contralateral pulmonary function with a chest radiograph and chest CT scan that do not show acute infiltrates
* FEV1 > or = to 2.0L on a preoperative pulmonary function test
* Karnofsky performance status of 70% or greater

Exclusion Criteria:

* Extended disease outside the ipsilateral hemithorax as determined by pre-operative radiographs or intraoperative findings
* Positive extrapleural nodes as determined by mediastinoscopy
* Positive LENIs
* Gross disease present within the hemithorax after surgery
* Evidence of distant metastases
* Severe non-malignant co-morbid disease: uncontrolled angina, myocardial infarction in the past 6 months, renal insufficiency, liver disease, pulmonary hypertension
* Presence of active concomitant malignancy
* Patients with a psychiatric or addictive disorder which would preclude informed consent
* Previous chemotherapy or radiation therapy to treat mesothelioma
* Chemotherapy or radiation therapy administered within 3 years for another malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2004-01; Primary Completion 2006-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To monitor tumor recurrence and patient survival, and compare those results to historic controls.

SECONDARY OUTCOMES:
To document the morbidity and mortality of this treatment protocol in this patient population | 3 years
to evaluate the pharmacokinetics of cisplatin. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: David J. Sugarbaker, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts